CLINICAL TRIAL: NCT00128167
Title: A Randomized, Double-Blind Trial to Assess the Safety and Relative Efficacy of CAIV-T Against Inactivated Influenza Vaccine in Children 6-59 Months of Age
Brief Title: Trivalent, Live, Cold Adapted Influenza Vaccine (CAIV-T) Against Inactivated Influenza Vaccine (TIV) in Children 6-59 Months of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: MI-CP111
Record Dates: First submitted 2005-08-05; First posted 2005-08-09 (Estimated); Last update posted 2021-09-13 (Actual); Status verified 2006-07

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

INTERVENTIONS:
Drug: Liquid CAIV-T

SUMMARY:
The primary objective of this study is to estimate the relative efficacy and assess the safety of CAIV-T compared to TIV.

ELIGIBILITY:
Inclusion Criteria:

* Age 6-59 months of age (not yet reached their 5th birthday)
* Parent or guardian available by telephone
* Available for illness visits at clinic or at home during the influenza surveillance period
* Written informed consent (and Health Insurance Portability and Accountability Act [HIPAA] authorization for U.S. Participants) obtained from the participant's parent or legal guardian and
* Ability of the parent/guardian to understand and comply with the requirements of the protocol

Exclusion Criteria:

* History of hypersensitivity to any component of CAIV-T or inactivated influenza vaccine, including egg or egg protein
* History of hypersensitivity to gentamicin
* Any known immunosuppressive condition or immune deficiency disease (including HIV infection), or ongoing receipt of any immunosuppressive therapy
* History of Guillain-Barre syndrome
* Medically-diagnosed wheezing, bronchodilator use, or steroid use (systemic or inhaled) within the previous 42 days by parent report or chart review (e.g., children with recent persistent asthma are excluded), or history of severe asthma
* Acute febrile (>100.0 degrees F or >37.8 degrees C oral or equivalent) illness or acute respiratory illness, including sore throat, within three days prior to enrollment
* Receipt of an investigational product within 30 days prior to enrollment or expected receipt during this study
* Use of aspirin or salicylate-containing products 30 days prior to enrollment or expected receipt during this study
* Use of anti-influenza medications (including amantadine, rimantadine, oseltamivir, and zanamivir) within 14 days prior to enrollment or expected receipt during this study
* Receipt of any blood product within 90 days prior to vaccination or expected receipt during this study
* Administration of any live virus vaccine within 30 days prior to enrollment, or if receipt of another live virus vaccine is expected within 30 days of any study vaccination
* Administration of any inactivated vaccine within 14 days prior to enrollment or if receipt of another inactivated vaccine is expected within 14 days prior to enrollment or if receipt of another inactivated vaccine is expected within 14 days of any study vaccination
* Close contact who is severely immunocompromised (e.g., transplant recipient)
* Family member or household contact who is an employee of the research center or otherwise involved with the conduct of the study and
* Any condition that, in the opinion of the investigator, might interfere with the interpretation or evaluation of the vaccines.

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 8500
Dates: Start 2004-10; Study Completion 2005-12

PRIMARY OUTCOMES:
The primary efficacy endpoint of this study is the relative efficacy of CAIV-T
compared to TIV against the incidence of culture-confirmed symptomatic influenza infection caused by community-acquired wild-type strains antigenically similar to those contained in the vaccine, occurring during the
influenza surveillance period and at least 14 days after the last required vaccination

SECONDARY OUTCOMES:
Culture-confirmed symptomatic influenza infection regardless of antigenic match
Febrile acute otitis media (AOM) with antibiotic use associated with culture-confirmed influenza infection antigenically similar to vaccine strains
Febrile acute otitis media (AOM) with antibiotic use associated with culture-confirmed influenza infection regardless of antigenic match
Lower respiratory illness (LRI) with culture-confirmed influenza infection antigenically similar to vaccine strains and
Lower respiratory illness (LRI) with culture-confirmed influenza infection regardless of antigenic match

CONTACTS AND LOCATIONS:
Overall Officials: Robert Walker, M.D., Study Director — MedImmune LLC
Locations (158):
- United States (107):
  - Clinical Research Consultants, Inc, Hoover, Alabama
  - University of Alabama, Tuscaloosa, Alabama
  - Little Rock Allergy and Asthma Clinical, Little Rock, Arkansas
  - Friendly Care Medical Group, Anaheim, California
  - Impact Clinical Trials, Beverly Hills, California
  - Family Medical Center, Foothill Ranch, California
  - Edinger Mecial Group, Fountain Valley, California
  - Fresno Childrens Medical Group, Inc., Fresno, California
  - Heathcare Partners Medical Group, Los Angeles, California
  - Kaiser Permanente Vaccine Study Center, Oakland, California
  - PRA Trials, Rolling Hills Estates, California
  - Benchmark Research, San Francisco, California
  - Convenience Care, West Covina, California
  - Norwich Pediatric Group, PC, Norwich, Connecticut
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Clinical Research Care & Resource Center, Inc, Miami, Florida
  - Suncoast Clinical Research, New Port Richey, Florida
  - Pediatric Research Center of South Florida, Palm Beach Gardens, Florida
  - Emory University School of Medicine, Dept of Pediatrics, Div of Infectious Diseases, Atlanta, Georgia
  - Pediatrics and Adolescent Medicine, P.A., Marietta, Georgia
  - Medical Parameters, Martinez, Georgia
  - Rush University Medical Center/University Consultatnts in Allergy and Immunology, Chicago, Illinois
  - Children's Memorial Hospital, Chicago, Illinois
  - Sneeze, Wheeze, & Itch Associates, LLC, Normal, Illinois
  - South Bend Clinic, South Bend, Indiana
  - Heart of America Research Institute, Shawnee Mission, Kansas
  - Heart of America Research Institute-Topeka, Topeka, Kansas
  - Kentucky Pediatrics/Adult Research Inc., Bardstown, Kentucky
  - University Child Health Specialists, PCTU, Louisville, Kentucky
  - Clinical Trials Management, LLC/The Pediatric Clinic, Bogalusa, Louisiana
  - Dolby Providers LLC, New Orleans, Louisiana
  - Boston University Medical Center, Boston, Massachusetts
  - Woburn Pediatric Associates, Woburn, Massachusetts
  - Odyssey Research, Dearborn, Michigan
  - Chidren's Hospital of Michigan, Detroit, Michigan
  - Center for Vaccine Development, St Louis, Missouri
  - Bozeman Urgent Care Center, Bozeman, Montana
  - Creighton/UNMC Pediatric Infectious Disease, Omaha, Nebraska
  - Meridian Clinical Research, LLC, Omaha, Nebraska
  - Henderson Pediatrics, Henderson, Nevada
  - Clinical Research Center of Nevada, Las Vegas, Nevada
  - Summit Pediatric Pulmonary, Summit, New Jersey
  - United Medical Associates, Binghamton, New York
  - Barbara Dzierzek/PharmaTrials, Inc., Brooklyn, New York
  - Health Sciences Research Center, Cortland, New York
  - Endwell Family Physicians, Endwell, New York
  - Winthrop University Hospital, Mineola, New York
  - Clarkstown Pediatric Associates, Nanuet, New York
  - CPMC Research Pharmacy, New York, New York
  - Elmwood Pediatrics, Rochester, New York
  - University Rochester Medical Center, Rochester, New York
  - Northeast Pediatrics and Adolescent Medicine, Syracuse, New York
  - Jacobi Medical Center, The Bronx, New York
  - Montefiore Medical Center, The Bronx, New York
  - Boone Pediatric Center, Boone, North Carolina
  - University of North Carolina Department of Pediatrics, Chapel Hill, North Carolina
  - Purcell Clinic, Laurinburg, North Carolina
  - North Carolina Clinical Research, Raleigh, North Carolina
  - Sylva Pediatrics Associates, Sylva, North Carolina
  - Ford, Simpson, Lively and Rice Pediatrics, Winston-Salem, North Carolina
  - Odyssey Research, Bismarck, North Dakota
  - Dakota Clinic/Innovis Health, Fargo, North Dakota
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Pediatric Associates of Mt. Carmel, Cincinnati, Ohio
  - Ohio Pediatrics, Huber Heights, Ohio
  - Shelly Senders and Associates, University Heights, Ohio
  - Grand Prairie Pediatric and Allergy Clinic, Oklahoma City, Oklahoma
  - Hillcrest Medical Group/Utica Park Clinic, Tulsa, Oklahoma
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Primary Physicians Research Inc., Pittsburgh, Pennsylvania
  - Asthma & Allergy Research Associates, Upland, Pennsylvania
  - East Bay Pediatrics, Barrington, Rhode Island
  - Omega Medical Research, Cranston, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Northridge Brown Clinic, Watertown, South Dakota
  - Medsouth Healthcare, Dyersburg, Tennessee
  - Holston Medical Group Pediatrics, Kingsport, Tennessee
  - Murfressboro Medical Clinic, Murfreesboro, Tennessee
  - Pediatric Clincal Research Office, Nashville, Tennessee
  - Wells Branch Medical Center, Austin, Texas
  - Sadler Clinic/Healthsouth Clinical Research, Conroe, Texas
  - Pediatric Allergy/Immunology Associates, PA, Dallas, Texas
  - Healthfirst Medical Group, Fort Worth, Texas
  - Med-Pro Research Inc., Houston, Texas
  - Scott and White/Pediatric Clinic, Killeen, Texas
  - Rd Clinical Research Inc., Lake Jackson, Texas
  - Central Texas Health Research, New Braunfels, Texas
  - Benchmark Research, San Angelo, Texas
  - Quality Assurance Research Center, San Antonio, Texas
  - Wee Care Pediatrics, Layton, Utah
  - Cottonwood Pediatrics, Murray, Utah
  - Bear Care Pediatrics, Ogden, Utah
  - Alpine Pediatrics, Pleasant Grove, Utah
  - Utah Valley Pediatrics, Provo, Utah
  - J. Lewis Research Inc., Salt Lake City, Utah
  - J. Lewis Research, Inc., Salt Lake City, Utah
  - Families First Pediatrics, South Jordan, Utah
  - J. Lewis Research/Southwest Family Medicine, West Jordan, Utah
  - PI-Coor Clinical Research, LLC, Burke, Virginia
  - Respiratory Disease Study Unit, Charlottesville, Virginia
  - Health Research of Hampton Roads, Inc, Newport News, Virginia
  - Center for Pediatric Research, Norfolk, Virginia
  - VCU Campus Children's Pavilion/Pediatric Clinical Trials Office, Richmond, Virginia
  - Advanced Pediatrics, Vienna, Virginia
  - Univeristy Pediatrics, Huntington, West Virginia
  - Monroe Medical Foundation, Monroe, Wisconsin
- Belgium (9):
  - Sint-Vincentiusziekenhuis Sint-Vincentiusstraat, Antwerp
  - Private Practice, Berchem
  - UVC Brugmann, Brussels
  - AZ-VUB Paediatric Clinic, Brussels
  - Private Practice, Drongen
  - KUL Dienst Jeugdgezondheidszorg, Leuven
  - Private Practice, Schoten
  - Private Practice, Tienen
  - Private Practice, Wondelgem
- Czechia (6):
  - IN Boskovice a. s. Detské oddelení, Boskovice
  - In Boskovice a.s. Detske oddeleni, Boskovice
  - Privantni praxe praktickenho, Lysice
  - Privátní praxe praktického lékare pro deti a dorost Lysice, Lysice
  - Nemocnice s poliklinikou v Moste, Most
  - STOPED s.r.o., Pilsen
- Hong Kong (5):
  - Department of Pediatrics, Chai Wan
  - Department of Pediatrics/Adolescent Medicine, Hang Hau
  - Department of Pediatrics - Paediatrics Unit, Kowloon
  - Department of Pediatrics/Adolescent Medicine, Lai Chi Kok
  - Department of Pediactrics, Shatin
- Ireland (3):
  - Springhill Surgery, Bangor County
  - Randalstown Health Centre, Randalsotown
  - Nottinghill Practice, Whiteabbey Health Centre, Whiteabbey
- South Korea (2):
  - Department of Pediatrics, Seoul
  - Dept. of Pediatrics, Seoul
- Taiwan (4):
  - Department of Pediatrics, Changhua
  - Department of Pediatrics, Taichung
  - Department of Pediatrics, Taipei
  - Department of Pediatrics, Taoyuan District
- United Kingdom (22):
  - Ashville Medical Center, Barnsely, South Yorks
  - Cathcart Street Practice, Ayr
  - Townhead Surgery, Ayrshire
  - Stonehill Medical Centre, Bolton
  - The Orchard Medical Centre, Bristol
  - The Staploe Medical Centre, Cambs
  - Avondale Surgery Research, Chesterfield
  - Saltash Health Centre, Cornwall
  - Woodend Health Centre, Coventry
  - Gabels Medical Centre, Coventry
  - Govind Health Cenre, Coventry
  - Woolwell Medical Centre, Devon Plymouth
  - The Medical Centre, East Horley
  - Valleyfield Health Centre, Fife
  - Castlemilk Health Centre, Glasgow
  - Kingsway Medical, Glasgow
  - Layton Medical Centre, Lancs
  - Greenwood & Sneinton Family Medical Practice, Nottingham
  - Landsdowne Road Yaxley, Peterborough
  - Knowle House Surgery, Plymouth
  - Wansford Surgery, Wansford
  - Sherbourne Medical Centre, Warwick Shire

REFERENCES:
- [Derived] Belshe RB, Edwards KM, Vesikari T, Black SV, Walker RE, Hultquist M, Kemble G, Connor EM; CAIV-T Comparative Efficacy Study Group. Live attenuated versus inactivated influenza vaccine in infants and young children. N Engl J Med. 2007 Feb 15;356(7):685-96. doi: 10.1056/NEJMoa065368. PMID 17301299